CLINICAL TRIAL: NCT02812563
Title: Familial Analysis of Keratoconus Risk
Acronym: AFRIK
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2013/03
Record Dates: First submitted 2015-07-07; First posted 2016-06-24 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: genetic — Galilee exam - Corn analysis with Optiwave Refractive Analysis

SUMMARY:
The principal objective of this study is to evaluate the frequency of KC inside family of patients with confirmed KC.

It's a familial, epidemiological, prospective, single-center study.

DETAILED DESCRIPTION:
Keratoconus is a common bilateral progressive corneal ectatic disease causing visual impairment by inducing irregular astigmatism and corneal opacities. This disorder typically begins during teenage years, progresses until the age of 30 to 40 years and, in severe forms, may need a corneal transplantation.

Currently, keratoconus has not known etiopathogenesis, and it is difficult to detect subclinical forms.

Several risk factors seem to be implied, environmental and genetic : the risk of keratoconus in case of familial history of keratoconus isn't well known at that time, but seems to be important to consider to promote screening and follow up of patient with a familial history of keratoconus (KC).

ELIGIBILITY:
Inclusion Criteria:

Case :

* patient carrier of keratoconus
* more than 7 years
* patient who didn't expressed opposition as for computerization and use of data concerning him

Family of case

* to have a first degree family member (father, mother, brother, sister, child) carrier of keratoconus
* more than 7 years
* patient who didn't expressed opposition as for computerization and use of data concerning him

Exclusion Criteria:

* ocular pathology or antecedent of modification of cornea (surgery, traumatism, ocular hypertension, keratitis) which could interfere with topographical analysis
* wearing of rigid contact lens for 15 days before exams, or flexible lens for 5 days before exams

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients + 2-5 members of family.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
proportion of diagnosed keratoconus | 1 day

SECONDARY OUTCOMES:
Assesment of familial history on KC severity | 1 day
Evaluation of KC severity | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: David Touboul, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Centre de Référence National du Kératocône Service d'ophtalmologie - Hôpital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Millodot M, Shneor E, Albou S, Atlani E, Gordon-Shaag A. Prevalence and associated factors of keratoconus in Jerusalem: a cross-sectional study. Ophthalmic Epidemiol. 2011 Apr;18(2):91-7. doi: 10.3109/09286586.2011.560747. PMID 21401417
- [Background] Weed KH, MacEwen CJ, Giles T, Low J, McGhee CN. The Dundee University Scottish Keratoconus study: demographics, corneal signs, associated diseases, and eye rubbing. Eye (Lond). 2008 Apr;22(4):534-41. doi: 10.1038/sj.eye.6702692. Epub 2007 Jan 19. PMID 17237755
- [Background] Assiri AA, Yousuf BI, Quantock AJ, Murphy PJ. Incidence and severity of keratoconus in Asir province, Saudi Arabia. Br J Ophthalmol. 2005 Nov;89(11):1403-6. doi: 10.1136/bjo.2005.074955. PMID 16234439
- [Background] Owens H, Gamble G. A profile of keratoconus in New Zealand. Cornea. 2003 Mar;22(2):122-5. doi: 10.1097/00003226-200303000-00008. PMID 12605045
- [Background] McMonnies CW, Boneham GC. Keratoconus, allergy, itch, eye-rubbing and hand-dominance. Clin Exp Optom. 2003 Nov;86(6):376-84. doi: 10.1111/j.1444-0938.2003.tb03082.x. PMID 14632614
- [Background] Falls HF, Allen AW. Dominantly inherited keratoconus. J Genet Hum. 1969 Oct;17(3):317-24. No abstract available. PMID 5387413
- [Background] Kemp EG, Lewis CJ. Measurement of total and specific IgE levels in the management of a family exhibiting a high incidence of keratoconus. Acta Ophthalmol (Copenh). 1984 Aug;62(4):524-9. doi: 10.1111/j.1755-3768.1984.tb03963.x. PMID 6485750
- [Background] Ihalainen A. Clinical and epidemiological features of keratoconus genetic and external factors in the pathogenesis of the disease. Acta Ophthalmol Suppl (1985). 1986;178:1-64. PMID 3019073
- [Background] Rabinowitz YS, Garbus J, McDonnell PJ. Computer-assisted corneal topography in family members of patients with keratoconus. Arch Ophthalmol. 1990 Mar;108(3):365-71. doi: 10.1001/archopht.1990.01070050063032. PMID 2310336